CLINICAL TRIAL: NCT00854620
Title: A Phase 2 Study of Sorafenib in Patients With Metastatic Renal Cell Carcinoma at Stanford University
Brief Title: Safety and Toxicity Study of Sorafenib in Patients With Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sandy Srinivas, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-04988; 96919 (Other: Stanford Secondary IRB Approval Number); SU-02272009-1898 (Other: Stanford University); RENAL0009 (Other: OnCore)
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Carcinoma, Renal Cell; Kidney Disease; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Diseases; Kidney Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): * Cycle 1: 400 mg BID sorafenib
  * Cycle 2: 600 mg BID sorafenib
  * Cycle 3+: 800 mg BID sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib administered in escalating 28-days cycles (400, 600 and 800 mg BID)
  Other Names: Nexavar; Sorafenib tosylate

SUMMARY:
Determine time-to-progression (TTP) for an escalating dose schedule for subjects with progressive metastatic renal cell carcinoma treated with sorafenib

DETAILED DESCRIPTION:
Sorafenib to be administered as 28-day cycles.

Sorafenib dose escalation by cycle is:

* Cycle 1: 400 mg BID
* Cycle 2: 600 mg BID
* Cycle 3+: 800 mg BID

Within subject dose escalation and maximum dose is dependent on observed tolerability.

Dose escalation only occurs after acceptable tolerability is demonstrated by subject.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- or cytologically-confirmed metastatic or unresectable renal cell carcinoma (RCC).
2. must have a component of conventional clear cell renal carcinoma.
3. No more than one prior systemic therapy.
4. No prior vascular endothelial growth factor receptor agents.
5. Prior palliative radiotherapy in metastatic lesion(s) is permitted, provided the subject has at least one measurable and/or evaluable lesion(s) that has not been irradiated.
6. All major surgery of any type and/or radiotherapy must be completed at least 4 weeks prior to Day 1 dosing. Patients must have recovered from surgery and/or radiotherapy toxicity prior to Day 1 dosing.
7. Measureable disease by RECIST criteria
8. Karnofsky performance status at least 70% or ECOG not more than 2
9. Ability to give written informed consent
10. At least 18 years old
11. Negative pregnancy test within 7 days of Day 1 dosing (female subjects of childbearing potential)
12. Sexually active fertile subjects must agree to use an accepted method of contraception during the course of the study for 3 months thereafter.
13. ANC at least 1,500/uL
14. Platelet count at least 100,000/uL
15. AST/ALT not more than 2.5 times the upper limit of normal (ULN)
16. Alkaline phosphatase not more than 2.5 x ULN
17. Serum bilirubin not more than 1.5 x ULN
18. Amylase/Lipase within normal range
19. Urinalysis not more than 1+ protein
20. Serum creatinine not more than 1.5 x ULN
21. No active ischemia by ECG
22. Echocardiogram or MUGA ejection fraction at least 40%

Exclusion Criteria:

1. Ongoing hemoptysis
2. Cerebrovascular accident within 12 months
3. Peripheral vascular disease with claudication on less than 1 block
4. History of clinically significant bleeding
5. Malignancy with true papillary/sarcomatoid features without any clear cell component
6. Chromophobe
7. Oncocytoma
8. Collecting duct tumors
9. Transitional cell carcinoma
10. Deep venous thrombosis or pulmonary embolus within one year of consent
11. Ongoing need for full-dose oral or parenteral anticoagulation. Low dose coumadin (1 mg) for maintenance of catheter patency or daily prophylactic aspirin is allowed
12. Subjects with evidence of current central nervous system (CNS) metastases
13. MRI or CT scan of the brain (with contrast, if possible) within 28 days prior to Day 1 dosing
14. Significant cardiovascular disease defined as congestive heart failure (New York Heart Association Class II, II or IV)
15. Angina pectoris requiring nitrate therapy
16. Myocardial infarction within the last 6 months
17. Uncontrolled hypertension (defined as blood pressure at least 160 mmHg systolic or at least 90 mmHg diastolic on medication)
18. Ongoing requirement for systemic corticosteroid therapy (except replacement therapy for adrenal insufficiency). Topical and/or inhaled steroids are allowed.
19. Uncontrolled psychiatric disorder
20. Delayed healing of wounds, ulcers, and/or bone fractures
21. Prior malignancy (EXCEPTIONS: adequately-treated basal cell or squamous cell skin cancer or any other cancer for which chemotherapy has been completed > 5 years ago and from which the patient has been disease-free for > 5 years)
22. Pregnant
23. Currently lactating
24. Currently using St John's Wort (an herb)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib: * Cycle 1: 400 mg BID sorafenib
  * Cycle 2: 600 mg BID sorafenib
  * Cycle 3+: 800 mg BID sorafenib
  Sorafenib: Sorafenib administered in escalating 28-days cycles (400, 600 and 800 mg BID)
Period: Overall Study
Arm/Group | Sorafenib
Started | 9
Completed | 8
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All subjects enrolled were included in the analysis
Arm/Group | Sorafenib
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 60 [47 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Time-to-progression (TTP)
Time Frame: 12 months
Measure: Median (Full Range); unit: months
Arm/Group | Sorafenib
Number analyzed (Participants) | 9
months | 5.3 [0.9 to 9.5]

ADVERSE EVENTS:
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (N=9)
General disorders and administration site conditions-other, Hand foot Syndrome (General disorders) | 9 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 9 (15)
Hypertension (Vascular disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (3)
Weight loss (Investigations) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No